CLINICAL TRIAL: NCT06018506
Title: A Phase I ,Single-arm, Open-label Study to Evalute the Safety, Tolerability, Pharmacokinetics, Immunogenicity, and Clinical Activity of BR108 Injection in Subjects With Hematological Malignancies
Brief Title: A Phase I Study of BR108 in Hematological Malignancies
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Adjustment of Company R&D strategy
Sponsor: BioRay Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BR108
Record Dates: First submitted 2023-08-11; First posted 2023-08-30 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-11

CONDITIONS: Hematologic Malignancy
MeSH Terms: conditions — Hematologic Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- BR108 (Experimental)
  Interventions: Drug: BR108 injection

INTERVENTIONS:
Drug: BR108 injection — Given into the vein (IV; intravenously) on Days 1 and 15 of each treatment cycle

SUMMARY:
A Phase I study of BR108 in hematological malignancies

ELIGIBILITY:
Inclusion Criteria:

* 1. Voluntary agreement to provide written informed consent;
* 2. Males and females who are ≥18 years old;
* 3. Patients must have an advanced hematologic malignancy including： Relapsed or refractory lymphoma as defined by World Health Organization(WHO) criteria； Relapsed or refractory AML /MDSas defined by World Health Organization (WHO) criteria；
* 4. Subjects must have documented CD70-positive .
* 5. Eastern Cooperative Oncology Group (ECOG) performance status of 0-2;
* 7. Expected survival time ≥3 months;
* 8.Have at least 1 evaluable lesion per Lugano 2014;
* 9. The function of major organs must meet the following criteria (Lymphoma：have not received blood transfusion, EPO, G-CSF or other medical supportive treatment within 7 days before the first dose of study drug) ：

  * White blood cell count≤25×109/L（for AML/MDS）
  * Absolute neutrophil count (ANC) ≥1.5×109/L or ≥0.75×109 /L for patients with bone marrow infiltration, Platelet ≥75×109 /L or ≥50×109 /L for patients with bone marrow infiltration; Hemoglobin ≥8.0mmol/L or ≥ 7.0mmol/L for patients with bone marrow infiltration;
  * International normalized ratio (INR) or prothrombin time (PT) ≤1.5×ULN; Activated Partial Thromboplastin Time (APTT) ≤1.5×ULN;
  * serum creatinine≤1.5×ULN or Creatinine clearance rate ≥60 mL/min ;
  * Total bilirubin ≤1.5×ULN or ≤3×ULN for patients with Gilbert's syndrome or liver metastasis； Aspartate aminotransferase (AST) and Alanine aminotransferase (ALT) ≤2.5×ULN or ≤5×ULN for patients with liver metastasis:
* 10. Women of child bearing potential and non-sterilized male patients who are sexually active with a female partner of child bearing potential must agree to use an effective method of contraception from screening until 6 months after the last dose of study drug. Effective methods of contraception consist of prior sterilization, intrauterine device, intrauterine hormone-releasing system, oral or injectable contraceptives, and sexual abstinence.
* 11. Patients will be able to communicate well with the investigator, understand and comply with the requirements of the study.

Exclusion Criteria:

* 1. Pregnant or lactating women;
* 2. Acute promyelocytic leukemia, acute transformation of chronic myeloid leukemia, primary central nervous system malignancies or invasion of the central nervous system (except for those who are asymptomatic or stable and do not require treatment ≥4 weeks before the first dose of study drug);
* 3. Has not recovered from adverse reactions caused by previous anti-tumor treatments to ≤ grade 1 or baseline (refer to NCICTCAE5.0 ), except for alopecia, pigmentation and other toxicity judged no safety risk by the investigator;
* 4. Previous exposure to CD70-targeted agents;
* 5. Patients with Allergic history or hypersensitivity reaction to any components of BR108 injection;
* 6. Patients with active bacterial, viral, fungal, mycobacterium, parasite or other infection (except fungal infection of nail bed) within 7 days prior to enrollment and requiring intravenous infusion therapy (except neoplastic fever);
* 7. Patients with inherited or acquired hemorrhagic diseases or severe coagulation abnormalities of clinical significance（ Such as diffuse intravascular coagulation (DIC) autoimmune hemolytic anemia, idiopathic thrombocytopenic purpura, sickle cell anemia, etc）;
* 8. HBsAg or HBcAb positive, and HBV DNA positive; HCVAb positive and HCV RNA positive; HIV positive; syphilis infection requiring systematic treatment ;
* 9. Subjects who have received live or attenuated vaccine within 4 weeks before the first administration or planned to receive live vaccine during the study period;
* 10. History of any other malignancies within 3 years (except for basal cell carcinoma of the skin, squamous cell carcinoma of the skin, superficial bladder cancer, localized prostate cancer, cervical carcinoma in situ, stage I ductal carcinoma in situ of the breast, and malignancies that have been cured (CR) within 2 years prior to initial administration and are currently considered stable by the investigator with minimal risk of recurrence);
* 11. Patients with serious cardiovascular and cerebrovascular diseases or other serious organic diseases, including but not limited to:

  * History of stroke 、intracranial hemorrhage 、unstable angina pectoris、 congestive heart failure (NYHA III-IV)、myocardial infarction、severe arrhythmias (e.g., persistent ventricular tachycardia, ventricular fibrillation) or congenital long QT syndrome within 6 months before enrollment.
  * Left ventricular ejection fraction （LVEF） < 50% in echocardiography (ECHO) or muti-gate detection scan (MUGA) .
  * Corrected QT interval prolongation >470ms.
  * Patients with interstitial lung disease, severe lung dysfunction, severe pulmonary fibrosis, or pulmonary infection requiring systematic treatment.
* 12. Subjects who have autoimmune disorders and need to rely on immunosuppressive therapy or receive systemic therapy with a dose of ≥20mg/day of prednisone or other equivalent hormones within 2 weeks before enrollment;
* 13. Patients have received other clinical trials within 4 weeks before the first dose of study drug;
* 14.Subjects who have major surgery or severe trauma within 4 weeks prior to initial dosing or plan to take major surgery during the trial period;
* 15. Treatment with prior anti-cancer therapy (including chemotherapy, endocrine therapy, targeted therapy, etc.) must have been terminated at last 28 days or 5 half-lives (whichever is shorter) before study enrolment,2 weeks for endocrine therapy and Chinese medicine treatment with anti-tumor indications or local palliative radiotherapy for bone metastasis and pain relief within 2 weeks.
* 16. Prior allogeneic hematopoietic stem cell or organ transplantation; recent Autologous hematopoietic stem cell transplantation（less than 3 months prior first dosing of study drug）;
* 17. Patients with any mental or cognitive impairment that may restrict the understanding and implementation of the informed consent;
* 18. Other serious, uncontrollable concomitant diseases that may affect protocol compliance or interfere with outcomes, or other serious or uncontrollable medical conditions that the investigator believes may put subjects at risk for participating in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2023-03-18 (Actual); Primary Completion 2024-05-27 (Actual); Study Completion 2024-06-21 (Actual)

PRIMARY OUTCOMES:
Number of Participants with Dose Limiting Toxicity (DLT) | up to 28 days
  Dose limiting toxicity
objective response rate（ORR） | up to approximately 3 years
  FOR lymphoma ，Objective Response Rate is defined as the percentage of patients with a complete response (CR) or partial response (PR). For AML, the proportion of participants who achieve a best response of CR, CRi, MLFS, or partial response (PR). For MDS, the proportion of participants who achieve a best response of CR, marrow CR, or PR.

SECONDARY OUTCOMES:
Cmax | up to approximately 3 years
  Cmax is the maximum observed concentration.
Tmax | up to approximately 3 years
  Time to maximum concentration attained
Incidence of antidrug antibodies (ADA) | up to approximately 3 years
  Percentage of patients producing detectable ADA
Duration of remission (DOR) | up to approximately 3 years
  To preliminarily evaluate DoR in patients with hematological malignancies

CONTACTS AND LOCATIONS:
Locations (1):
- Tianjin Medical University Cancer Institute and Hospital, Tianjin, Tianjin Municipality, China

IPD SHARING:
Plan to Share IPD: No